CLINICAL TRIAL: NCT00265382
Title: 26-Week Open-Label Extension Study Evaluating The Safety And Tolerability Of Flexible Doses Of Oral Ziprasidone In Adolescent Subjects With Schizophrenia
Brief Title: Safety And Tolerability Of Ziprasidone In Adolescents With Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281135
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2010-05-19 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia
Keywords: Adolescent Subjects
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open (Other)
  Interventions: Drug: Ziprasidone oral capsules

INTERVENTIONS:
Drug: Ziprasidone oral capsules — Study medications will include oral ziprasidone capsules of 20 mg, 40 mg, 60 mg, and 80 mg strength. Subjects will be dosed daily for 26 weeks using a flexible dose design with a minimal dose range of 20mg bid to a maximum dose range of 80 mg bid.
  Other Names: Geodon, Zeldox

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ziprasidone during long-term open-label administration in adolescents (ages 13-17) with schizophrenia.

DETAILED DESCRIPTION:
On March 24, 2009, Pfizer Inc. stopped late stage Geodon pediatric clinical trials in schizophrenia (A1281134 - placebo controlled; A1281135 - open label). As recommended by the DSMB, these studies were stopped due to lack of efficacy. No safety concerns were identified.

ELIGIBILITY:
Inclusion Criteria:

* Participation in double-blind treatment study A1281134, meeting specific criteria of duration and safety

Exclusion Criteria:

* Imminent risk of suicide or homicide, as judged by the site investigator
* Serious adverse event related to study medication in study A1281134
* Significant prolongation of QT interval in study A1281134

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (21):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Altamonte Springs, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Smyrna, Georgia
  - Pfizer Investigational Site, Tucker, Georgia
  - Pfizer Investigational Site, Des Plaines, Illinois
  - Pfizer Investigational Site, Oakbrook Terrace, Illinois
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Clinton Township, Michigan
  - Pfizer Investigational Site, Bridgeton, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Bothell, Washington
  - Pfizer Investigational Site, Spokane, Washington
- Colombia (2):
  - Pfizer Investigational Site, Bello, Antioquia
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Pfizer Investigational Site, San José, Costa Rica
- India (8):
  - Pfizer Investigational Site, Vijaywada, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Guj
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Aurangabad, Maharashtra
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Chennai, Tamil Nadu
- Malaysia (2):
  - Pfizer Investigational Site, Kubang Kerian, Kelantan
  - Pfizer Investigational Site, Kuala Lumpur
- Pfizer Investigational Site, Lima, Peru
- Russia (7):
  - Pfizer Investigational Site, Lipetsk Region, Russia
  - Pfizer Investigational Site, Kazan'
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Nizhny Novgorod
  - Pfizer Investigational Site, Saratov
  - Pfizer Investigational Site, Tver'
  - Pfizer Investigational Site, Yaroslavl
- Pfizer Investigational Site, Singapore, Singapore
- Ukraine (10):
  - Pfizer Investigational Site, Simferopol, Autonomous Republic of Crimea
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Luhansk
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Odesa
  - Pfizer Investigational Site, Poltava
  - Pfizer Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Findling RL, Cavus I, Pappadopulos E, Vanderburg DG, Schwartz JH, Gundapaneni BK, DelBello MP. Ziprasidone in adolescents with schizophrenia: results from a placebo-controlled efficacy and long-term open-extension study. J Child Adolesc Psychopharmacol. 2013 Oct;23(8):531-44. doi: 10.1089/cap.2012.0068. Epub 2013 Oct 10. PMID 24111983
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281135&StudyName=Safety%20And%20Tolerability%20Of%20Ziprasidone%20In%20Adolescents%20With%20Schizophrenia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adolescent subjects with schizophrenia, ages 13-17 years, who participated in the double-blind placebo controlled Study A1281134 (NCT00257192) who met qualification criteria and wished to receive treatment with open-label ziprasidone.
Groups:
- Ziprasidone: Titrated over a 2-week period, starting with an evening dose of 20 milligrams (mg)/day, and subsequent dose increases of 20 mg/day every second day up to a target dose of 80 to 160 mg/day for subjects weighing > = 45 kilograms (kg). For subjects with a body weight < 45 kg, the maximum permitted dose was 80 mg/day (40 mg twice a day [BID]). Doses could have been reduced to a minimum of 40 mg/day (20 mg BID).
Period: Overall Study
Arm/Group | Ziprasidone
Started | 221
Completed | 76
Not Completed | 145
Not completed — Adverse Event | 21
Not completed — Laboratory Abnormality | 1
Not completed — Lost to Follow-up | 3
Not completed — Lack of Efficacy | 6
Not completed — Miscellaneous | 6
Not completed — Withdrawal by Subject | 13
Not completed — Study terminated by sponsor | 94
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Ziprasidone: Titrated over a 2-week period, starting with an evening dose of 20 mg/day, and subsequent dose increases of 20 mg/day every second day up to a target dose of 80 to 160 mg/day for subjects weighing > = 45 kg. For subjects with a body weight < 45 kg, the maximum permitted dose was 80 mg/day (40 mg BID). Doses could have been reduced to a minimum of 40 mg/day (20 mg BID).
Arm/Group | Ziprasidone
Number analyzed (Participants) | 221
Age, Customized [Number; unit: Participants] — Baseline data are from the preceding Study A1281134 (NCT00257192).
  Participants
    >12 years and <13 years at start of treatment | 3
    13 to 17 years | 218
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: All observed or volunteered treatment-emergent AEs and SAEs regardless of treatment group or suspected causal relationship to the investigational product(s) were reported.
Time Frame: 26 weeks
Population: Safety Analysis Set = all subjects who took at least one dose of study medication. In this table, the number of subjects with AEs is based on a 0% AE threshold whereas the number of subjects with AEs reported in the AE section are based on a 5% AE threshold.
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 221
participants
  AEs | 137
  SAEs | 16

2. Secondary Outcome: Number of Subjects With Change From Baseline to Each Pubertal Stage of Development as Assessed by the Tanner Adolescent Pubertal Self Assessment
Description: Tanner Adolescent Pubertal Staging Questionnaire: used to document the stage of development of secondary sexual characteristics. Female pubertal development staged by pubic hair development and breast size; males pubertal development staged by size of the genitalia and development of pubic hair. Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size).
Time Frame: Baseline, Week 26, Early Termination (ET)
Population: Safety Analysis Set. N=number of subjects with analyzable data at baseline. Baseline data from Study A1281134 (NCT00257192) served as the baseline for A1281135.
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 73
participants
  Pubic Hair, Week 26 (Stage 1) | 1
  Pubic Hair, Week 26 (Stage 2) | 1
  Pubic Hair, Week 26 (Stage 3) | 11
  Pubic Hair, Week 26 (Stage 4) | 39
  Pubic Hair, Week 26 (Stage 5) | 21
  Pubic Hair, ET (Stage 1) | 0
  Pubic Hair, ET (Stage 2) | 10
  Pubic Hair, ET (Stage 3) | 22
  Pubic Hair, ET (Stage 4) | 59
  Pubic Hair, ET (Stage 5) | 30

3. Secondary Outcome: Change From Baseline in Children's Problem Behavior and Aggression Questionnaire (CPBAQ) Total Score
Description: CPBAQ: 19-item parent or legal guardian completed questionnaire to rate the child's verbal (such as yelling or cursing) and physical aggression (such a fighting with peers or being cruel to an animal) during the past week. Behavior was rated on a 4-point scale; range 0 (behavior did not occur or was not a problem) to 3 (behavior occurred a lot or was severe problem). Total score range 0 to 57; higher scores indicate a greater frequency and severity of aggression.
Time Frame: Baseline, Weeks 2, 6, 18, 26, ET
Population: Safety Analysis Set. N=number of subjects with analyzable data at baseline; n=number of subjects with analyzable data at post-baseline observation. Baseline was the last available observation from Study A1281134 (NCT00257192). Last Observation Carried Forward (LOCF) imputation used for Week 26 LOCF time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 208
scores on a scale
  Week 2 (n=178) | -0.3 (4.8)
  Week 6 (n=153) | -0.8 (6.1)
  Week 18 (n=93) | -0.5 (6.5)
  Week 26 (n=68) | 0.7 (7.7)
  ET (n=113) | 0.5 (7.1)
  Week 26 LOCF (n=177) | -0.5 (7.0)

4. Secondary Outcome: Change From Baseline in Child Depression Rating Scale - Revised (CDRS-R): Total Score
Description: CDRS-R: clinician-rated interview-based scale (with both child and parent or guardian) to assess 17 distinct symptom areas to derive an index of depression severity. Discrepancies between informants' responses were resolved by using most impaired rating given by valid informant. Rated on a 7-point scale; range from 1 (no impairment) to 7 (indicates greater impairment). Total score calculated as sum of the 17 items (range 1 to 119); higher score indicates greater impairment.
Time Frame: Baseline, Weeks 1, 2, 6, 10, 14, 18, 22, 26, ET
Population: Safety Analysis Set. N=number of subjects with analyzable data at baseline; n=number of subjects with analyzable data at post-baseline observation. Baseline was the last available observation from Study A1281134 (NCT00257192). LOCF imputation used for Week 26 LOCF time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 214
scores on a scale
  Week 1 (n=198) | -1.4 (4.8)
  Week 2 (n=188) | -2.2 (6.1)
  Week 6 (n=160) | -3.5 (6.3)
  Week 10 (n=129) | -4.6 (7.3)
  Week 14 (n=105) | -5.0 (7.4)
  Week 18 (n=94) | -4.9 (8.1)
  Week 22 (n=78) | -5.1 (7.9)
  Week 26 (n=72) | -5.3 (7.8)
  ET (n=122) | -2.7 (7.3)
  Week 26 LOCF (n=197) | -4.5 (7.0)

5. Secondary Outcome: Change From Baseline in CNS Vital Signs Cognitive Test Battery (Includes Sedation Item): Subscales
Description: Computerized subject-administered test battery with subtests for verbal and visual memory, processing speed, nonverbal reasoning, executive functioning, working memory, sustained attention. Computerized 7- point sedation item (0 [not sleepy] to 10 [very sleepy]) was completed prior to test battery. Neurocognitive index score was derived from subtest scores per an algorithm. Index score and subtest scores assessed the subject's changes in cognition. Scores were rated as above average (score >109), average (90 to 109), below average (80 to 89), or well below average (70 to 79).
Time Frame: Baseline, Weeks 6 and 26, ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 212
scores on a scale
  Sedation: Week 6 (n=149) | 0.1 (1.7)
  Sedation: Week 26 (n=70) | -0.2 (1.5)
  Sedation: ET (n=102) | -0.1 (2.0)
  Sedation: Week 26 LOCF (n=153) | -0.2 (1.7)
  Verbal Memory: Week 6 (n=150) | -1.3 (13.7)
  Verbal Memory: Week 26 (n=71) | 0.6 (14.0)
  Verbal Memory: ET (n=103) | -0.7 (14.6)
  Verbal Memory: Week 26 LOCF (n=155) | 0.3 (14.5)
  Visual Memory: Week 6 (n=148) | -3.6 (13.7)
  Visual Memory: Week 26 (n=71) | -2.1 (15.5)
  Visual Memory: ET (n=103) | -1.9 (12.7)
  Visual Memory: Week 26 LOCF (n=154) | -1.5 (14.4)
  Processing Speed: Week 6 (n=148) | -1.2 (11.4)
  Processing Speed: Week 26 (n=71) | 2.1 (10.2)
  Processing Speed: ET (n=103) | -1.4 (19.0)
  Processing Speed: Week 26 LOCF (n=153) | 0.5 (12.0)
  Reasoning: Week 6 (n=145) | -0.3 (14.1)
  Reasoning: Week 26 (n=71) | 3.0 (11.3)
  Reasoning: ET (n=100) | 1.9 (14.9)
  Reasoning: Week 26 LOCF (n=151) | 1.5 (14.3)
  Executive Functioning: Week 6 (n=145) | 2.0 (16.7)
  Executive Functioning: Week 26 (n=71) | 2.0 (16.8)
  Executive Functioning: ET (n=100) | 2.4 (15.7)
  Executive Functioning: Week 26 LOCF (n=151) | 2.4 (16.9)
  Working Memory: Week 6 (n=145) | -0.5 (12.6)
  Working Memory: Week 26 (n=68) | 0.8 (16.4)
  Working Memory: ET (n=99) | 0.3 (12.1)
  Working Memory: Week 26 LOCF (n=150) | 0.7 (14.2)
  Sustained Attention: Week 6 (n=145) | 0.2 (12.0)
  Sustained Attention: Week 26 (n=68) | 1.9 (14.0)
  Sustained Attention: ET (n=99) | -0.6 (12.2)
  Sustained Attention: Week 26 LOCF (n=150) | 1.2 (12.7)

6. Secondary Outcome: Change From Baseline in CNS Vital Signs Cognitive Test Battery: Neurocognitive Index
Description: as for outcome 5
Time Frame: Baseline, Weeks 6 and 26, ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 208
scores on a scale
  Neurocognitive Index: Week 6 (n=144) | -0.6 (7.2)
  Neurocognitive Index: Week 26 (n=68) | 1.3 (7.3)
  Neurocognitive Index: ET (n=99) | 0.5 (6.3)
  Neurocognitive Index: Week 26 LOCF (n=150) | 0.7 (7.7)

7. Secondary Outcome: Change From Baseline in Simpson-Angus Rating Scale (SARS)
Description: SARS: 10-item clinician rated instrument to assess parkinsonian symptoms (7 items) and related extrapyramidal side effects (3 items): gait, arm dropping, shoulder shaking, elbow rigidity, leg pendulousness, glabellar tap, tremor, and salivation. Head dropping (modified SARS item 7) substituted for head rotation. Anchored 5-point scale: range 0 (absence of condition, normal) to 4 (most extreme form of condition). Total score is sum of individual item scores (range 0 to 40); higher score indicates more affected.
Time Frame: Baseline, Weeks 1, 2, 6, 10, 14, 18, 22, 26, ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 221
scores on a scale
  Week 1 (n=206) | -0.05 (1.4)
  Week 2 (n=197) | -0.11 (1.3)
  Week 6 (n=168) | -0.04 (1.7)
  Week 10 (n=135) | -0.10 (1.6)
  Week 14 (n=110) | -0.02 (1.9)
  Week 18 (n=99) | 0.02 (1.4)
  Week 22 (n=82) | -0.04 (1.7)
  Week 26 (n=76) | -0.32 (1.4)
  ET (n=127) | -0.31 (2.0)
  Week 26 LOCF (n=206) | -0.15 (1.5)

8. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BAS) Global Clinical Assessment Item
Description: BAS: clinician rated scale to assess akathisia to determine the degree of subjective restlessness and distress associated with restlessness. First 3 items (Objective, Subjective, and Distress related to restlessness) rated on a 4-point scale with range 0 (no symptoms) to 3 (increased severity of symptoms). Item 4 Global Clinical Assessment of Akathisia rated on a 6- point scale range 0 (no symptoms) to 5 (increased severity of symptoms); higher score indicates increased severity. All rating are anchored. Only the Global Clinical Assessment of Akathisia was to be analyzed.
Time Frame: Baseline, Weeks 1, 2, 6, 10, 14, 18, 22, 26, ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 221
scores on a scale
  Week 1 (n=206) | 0.0 (0.4)
  Week 2 (n=197) | 0.0 (0.4)
  Week 6 (n=168) | 0.0 (0.4)
  Week 10 (n=135) | 0.0 (0.5)
  Week 14 (n=110) | 0.1 (0.6)
  Week 18 (n=99) | 0.0 (0.4)
  Week 22 (n=82) | 0.0 (0.6)
  Week 26 (n=76) | 0.0 (0.6)
  ET (n=127) | 0.0 (0.5)
  Week 26 LOCF (n=206) | 0.1 (0.5)

9. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Movement Cluster Score
Description: AIMS: clinician rated 12-item scale to rate 7 body areas and global judgments on the severity of abnormal movements, incapacitation and subject's awareness of abnormal movements. Items 1 to 10 scored 0 (none) to 4 (severe) (total possible score 0 to 40; higher score indicates greater severity); items 11 to 14 are No or Yes response to dental status and sleep movements. Only the sum of the first 7 items to be analyzed (AIMS Movement Cluster score). Total score 0 to 28; higher score indicates greater severity.
Time Frame: Baseline, Weeks 1, 2, 6, 10, 14, 18, 22, 26, ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 221
scores on a scale
  Week 1 (n=206) | 0.06 (1.3)
  Week 2 (n=197) | -0.05 (0.7)
  Week 6 (n=168) | -0.04 (0.9)
  Week 10 (n=135) | 0.02 (1.4)
  Week 14 (n=110) | 0.01 (0.9)
  Week 18 (n=99) | 0.01 (0.6)
  Week 22 (n=82) | 0.10 (1.2)
  Week 26 (n=76) | 0.08 (1.2)
  ET (n=127) | -0.12 (1.5)
  Week 26 LOCF (n=206) | 0.00 (1.0)

10. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale - Anchored (BPRS-A) Total Score
Description: BPRS-A: 18-item clinician rated scale to assess somatic concern, anxiety, emotional withdrawal, disorganization, hallucinatory behavior, guilt feelings, suspiciousness, disorientation, tension, mannerisms, posturing, grandiosity, depressive mood, hostility, motor retardation, uncooperativeness, unusual thought content, blunted affect, excitement. Ratings anchored to improve consistency for single rater over time or between raters. Items rated on 7-point scale 0 (not present) to 6 (extremely severe). Total score=sum of items (range 0 to 108); higher scores indicate increased pathology.
Time Frame: Baseline, Weeks 2, 6, 18, 26, ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 220
scores on a scale
  Week 2 (n=196) | -3.8 (7.8)
  Week 6 (n=167) | -6.1 (8.8)
  Week 18 (n=98) | -7.8 (11.0)
  Week 26 (n=75) | -8.5 (9.9)
  ET (n=127) | -4.0 (9.1)
  Week 26 LOCF (n=196) | -6.9 (8.9)

11. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS)
Description: CGAS: clinician-rated global assessment item for children based on symptoms and social functioning in home, school, and community settings. Scores on this single item range from 1 to 100 (higher levels indicate greater health) with descriptive anchors for every 10-point interval. Scores above 70 on this scale are considered within the "normal" range; lower score indicates need for increased supervision.
Time Frame: Baseline, Weeks 2, 6, 18, 26, ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 221
scores on a scale
  Week 2 (n=197) | 55.5 (12.9)
  Week 6 (n=168) | 59.2 (12.5)
  Week 18 (n=99) | 62.3 (11.4)
  Week 26 (n=76) | 65.6 (12.4)
  ET (n=127) | 56.6 (15.1)
  Week 26 LOCF (n=197) | 60.5 (14.2)

12. Secondary Outcome: Change From Baseline in Child Health Questionnaire (CHQ)
Description: CHQ: 50-item, 15 subscale parent or legal guardian assessed instrument of child's physical, emotional, social well-being, and relative burden of disease on the parents; rated on Likert-type scale: range 0 to 100; higher scores indicate a more positive health status. Global indicators for Physical Health and Psychosocial Health are weighted composites derived from subscale items using scoring algorithms (transformed scores); range 0 to 100: higher scores indicate more positive health status.
Time Frame: Baseline, Weeks 6 and 26, ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 220
scores on a scale
  Global Health: Week 6 (n=163) | 44.2 (23.9)
  Global Health: Week 26 (n=75) | 50.3 (22.1)
  Global Health: ET (n=124) | 40.5 (25.8)
  Global Health: Week 26 LOCF (n=164) | 44.9 (22.9)
  Global Behavior: Week 6 (n=163) | 44.9 (23.6)
  Global Behavior: Week 26 (n=75) | 47.0 (24.2)
  Global Behavior: ET (n=124) | 38.7 (25.8)
  Global Behavior: Week 26 LOCF (n=164) | 43.8 (24.4)
  Family Cohesion: Week 6 (n=163) | 53.0 (23.9)
  Family Cohesion: Week 26 (n=75) | 54.4 (24.7)
  Family Cohesion: ET (n=124) | 50.0 (23.9)
  Family Cohesion: Week 26 LOCF (n=164) | 53.4 (23.7)
  Physical Health: Week 6 (n=163) | 76.4 (30.8)
  Physical Health: Week 26 (n=74) | 80.2 (28.8)
  Physical Health: ET (n=123) | 75.5 (32.8)
  Physical Health: Week 26 LOCF (n=163) | 77.8 (31.2)
  Bodily Pain: Week 6 (n=163) | 80.8 (21.6)
  Bodily Pain: Week 26 (n=75) | 84.4 (21.5)
  Bodily Pain: ET (n=124) | 81.0 (22.7)
  Bodily Pain: Week 26 LOCF (n=164) | 82.5 (21.3)
  Emotion, Behavior: Week 6 (n=163) | 53.3 (32.6)
  Emotion, Behavior: Week 26 (n=74) | 60.1 (31.2)
  Emotion, Behavior: ET (n=123) | 49.5 (34.5)
  Emotion, Behavior: Week 26 LOCF (n=163) | 54.8 (32.2)
  Time Impact on Parent: Week 6 (n=163) | 62.0 (26.6)
  Time Impact on Parent: Week 26 (n=75) | 69.9 (23.5)
  Time Impact on Parent: ET (n=124) | 59.9 (28.6)
  Time Impact on Parent: Week 26 LOCF (n=164) | 65.1 (26.3)
  Emotional Impact on Parent: Week 6 (n=163) | 49.5 (24.6)
  Emotional Impact on Parent: Week 26 (n=75) | 57.2 (24.7)
  Emotional Impact on Parent: ET (n=124) | 43.4 (25.9)
  Emotional Impact on Parent: Week 26 LOCF (n=164) | 52.2 (26.0)
  Mental Health: Week 6 (n=163) | 63.6 (16.1)
  Mental Health: Week 26 (n=75) | 66.7 (16.5)
  Mental Health: ET (n=124) | 60.8 (18.3)
  Mental Health: Week 26 LOCF (n=164) | 65.1 (16.1)
  Physical Function: Week 6 (n=163) | 80.4 (22.3)
  Physical Function: Week 26 (n=75) | 84.9 (19.0)
  Physical Function: ET (n=124) | 79.5 (23.4)
  Physical Function: Week 26 LOCF (n=164) | 81.4 (21.9)
  Behavior Scale: Week 6 (n=163) | 62.7 (16.8)
  Behavior Scale: Week 26 (n=75) | 64.5 (20.0)
  Behavior Scale: ET (n=124) | 60.2 (18.7)
  Behavior Scale: Week 26 LOCF (n=164) | 63.0 (18.4)
  Self-Esteem: Week 6 (n=163) | 52.7 (20.3)
  Self-Esteem: Week 26 (n=74) | 55.3 (21.0)
  Self-Esteem: ET (n=124) | 52.6 (21.7)
  Self-Esteem: Week 26 LOCF (n=163) | 54.5 (20.6)
  General Health Perception: Week 6 (n=163) | 50.3 (15.3)
  General Health Perception: Week 26 (n=75) | 51.8 (16.4)
  General Health Perception: ET (n=124) | 49.7 (15.1)
  General Health Perception: Week 26 LOCF (n=164) | 50.3 (15.4)
  Family Activities: Week 6 (n=163) | 60.1 (24.9)
  Family Activities: Week 26 (n=75) | 63.9 (24.1)
  Family Activities: ET (n=124) | 56.3 (27.6)
  Family Activities: Week 26 LOCF (n=164) | 61.6 (26.1)
  Physical Health Global Subscale: Week 6 (n=163) | 44.1 (11.7)
  Physical Health Global Subscale: Week 26 (n=74) | 46.6 (10.9)
  Physical Health Global: ET (n=123) | 43.8 (12.9)
  Physical Health Global: Week 26 LOCF (n=163) | 44.8 (12.2)
  Psychosocial Health Global: Week 6 (n=163) | 35.7 (10.4)
  Psychosocial Health Global: Week 26 (n=74) | 38.5 (10.9)
  Psychosocial Health Global: ET (n=123) | 33.7 (11.9)
  Psychosocial Health Global: Week 26 LOCF (n=163) | 36.8 (10.7)

13. Secondary Outcome: Number of Subjects Per Response on the School Placement Questionnaire: School Situation
Description: School placement questionnaire: parent or legal guardian assessed questionnaire to determine whether the child is currently enrolled in school (or planned to be enrolled if on school holiday like summer break), whether attending regularly if enrolled, and how well the child is doing overall in school. Questions were modified from those used in the National Institute of Mental Health (NIMH) funded Treatment of Early Onset Schizophrenia Spectrum (TEOSS) study. Results determine whether subjects are currently attending school and qualitatively describe how well they are doing in school.
Time Frame: Baseline, Weeks 6 and 26, ET
Population: Safety Analysis Set. N=number of subjects analyzable for School Placement Questionnaire; n=number of subjects with analyzable data at baseline and post-baseline observation. Baseline was the last available observation from Study A1281134 (NCT00257192). LOCF imputation used for Week 26 LOCF time point.
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 221
participants
  Baseline: Enrolled or Attend (n=221) | 63
  Baseline: Not Attend or Mental Illness (n=221) | 59
  Baseline: Not Attend or Other (n=221) | 4
  Baseline: Enrolled or Vacation (n=221) | 26
  Baseline: Not Enrolled or Mental Illness (n=221) | 42
  Baseline: Not Enrolled or Other (n=221) | 27
  Week 6: Enrolled or Attend (n=166) | 68
  Week 6: Not Attend or Mental Illness (n=166) | 32
  Week 6: Not Attend or Other (n=166) | 1
  Week 6: Enrolled or Vacation (n=166) | 14
  Week 6: Not Enrolled or Mental Illness (n=166) | 29
  Week 6: Not Enrolled or Other (n=166) | 22
  Week 26: Enrolled or Attend (n=75) | 35
  Week 26: Not Attend or Mental Illness (n=75) | 9
  Week 26: Not Attend or Other (n=75) | 0
  Week 26: Enrolled or Vacation (n=75) | 5
  Week 26: Not Enrolled or Mental Illness (n=75) | 13
  Week 26: Not Enrolled or Other (n=75) | 13
  ET: Enrolled or Attend (n=125) | 42
  ET: Not Attend or Mental Illness (n=125) | 35
  ET: Not Attend or Other (n=125) | 1
  ET: Enrolled or Vacation (n=125) | 9
  ET: Not Enrolled or Mental Illness (n=125) | 21
  ET: Not Enrolled or Other (n=125) | 17
  Week 26 LOCF: Enrolled or Attend (n=166) | 75
  Week 26 LOCF: Not Attend or Mental Illness (n=166) | 30
  Week 26 LOCF: Not Attend or Other (n=166) | 1
  Week 26 LOCF: Enrolled or Vacation (n=166) | 8
  Wk 26 LOCF: Not Enrolled or Mental Illness (n=166) | 28
  Week 26 LOCF: Not Enrolled or Other (n=166) | 24

14. Secondary Outcome: Number of Subjects Per Response on the School Placement Questionnaire: School Attendance
Description: as for outcome 13
Time Frame: Baseline, Weeks 6 and 26, ET
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 133
participants
  Baseline: No Absences (n=133) | 25
  Baseline: Only a Few Absences (n=133) | 37
  Baseline: Frequent Absences (n=133) | 12
  Baseline: Did Not Attend (n=133) | 36
  Baseline: Not Applicable or Vacation (n=133) | 23
  Week 6: No Absences (n=95) | 31
  Week 6: Only a Few Absences (n=95) | 29
  Week 6: Frequent Absences (n=95) | 11
  Week 6: Did Not Attend (n=95) | 10
  Week 6: Not Applicable or Vacation (n=95) | 14
  Week 26: No Absences (n=42) | 14
  Week 26: Only a Few Absences (n=42) | 16
  Week 26: Frequent Absences (n=42) | 7
  Week 26: Did Not Attend (n=42) | 0
  Week 26: Not Applicable or Vacation (n=42) | 5
  ET: No Absences (n=62) | 16
  ET: Only a Few Absences (n=62) | 23
  ET: Frequent Absences (n=62) | 5
  ET: Did Not Attend (n=62) | 11
  ET: Not Applicable or Vacation (n=62) | 7
  Week 26 LOCF: No Absences (n=93) | 32
  Week 26 LOCF: Only a Few Absences (n=93) | 32
  Week 26 LOCF: Frequent Absences (n=93) | 14
  Week 26 LOCF: Did Not Attend (n=93) | 7
  Week 26 LOCF: Not Applicable or Vacation (n=93) | 8

15. Secondary Outcome: Number of Subjects Per Response on the School Placement Questionnaire: Overall School Performance
Description: as for outcome 13
Time Frame: Baseline, Weeks 6 and 26, ET
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 103
participants
  Baseline: Excellent (n=103) | 5
  Baseline: Good (n=103) | 25
  Baseline: Fair (n=103) | 40
  Baseline: Poor (n=103) | 23
  Baseline: Very Poor (n=103) | 10
  Week 6: Excellent (n=73) | 2
  Week 6: Good (n=73) | 23
  Week 6: Fair (n=73) | 34
  Week 6: Poor (n=73) | 14
  Week 6: Very Poor (n=73) | 0
  Week 26: Excellent (n=37) | 1
  Week 26: Good (n=37) | 10
  Week 26: Fair (n=37) | 18
  Week 26: Poor (n=37) | 5
  Week 26: Very Poor (n=37) | 3
  ET: Excellent (n=48) | 0
  ET: Good (n=48) | 15
  ET: Fair (n=48) | 23
  ET: Poor (n=48) | 6
  ET: Very Poor (n=48) | 4
  Week 26 LOCF: Excellent (n=80) | 1
  Week 26 LOCF: Good (n=80) | 22
  Week 26 LOCF: Fair (n=80) | 39
  Week 26 LOCF: Poor (n=80) | 15
  Week 26 LOCF: Very Poor (n=80) | 3

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are reported from time of first dose of study treatment up to 6 days after last dose of study treatment.
Description: Safety population = all randomized subjects with at least 1 dose of study treatment. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 16/221
Other Adverse Events (participants affected / at risk) | 68/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=221)
Drug ineffective (General disorders) | 1
Dystonia (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Delusional perception (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 2
Intentional self-injury (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 2
Persecutory delusion (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 4
Schizophrenia, paranoid type (Psychiatric disorders) | 1
Self injurious behaviour (Psychiatric disorders) | 2
Suicidal behaviour (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 3
Thinking abnormal (Psychiatric disorders) | 1
Sexual activity increased (Social circumstances) | 1
Victim of sexual abuse (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=221)
Headache (Nervous system disorders) | 20
Somnolence (Nervous system disorders) | 33
Tremor (Nervous system disorders) | 14
Fatigue (General disorders) | 11
Insomnia (Psychiatric disorders) | 11

LIMITATIONS AND CAVEATS:
The AE tables were amended to incorporate previously unreported AEs that were found during an independent audit and verified by the investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.